CLINICAL TRIAL: NCT04734236
Title: Development of a Rapid and Accurate Diagnostic Assay for Tuberculosis by Using New Sample Preparation and Detection Technique
Brief Title: Development of Molecular Diagnostic Platform for Tuberculosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, Dr, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RapidassaytestforTB
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New technique group (Active Comparator)
  Interventions: Diagnostic Test: New technique vs Xpert
- Xpert group (Sham Comparator)
  Interventions: Diagnostic Test: New technique vs Xpert

INTERVENTIONS:
Diagnostic Test: New technique vs Xpert — New technique vs Xpert

SUMMARY:
This study evaluates new technique for diagnosis of tuberculosis. Among patients who are suspected with tuberculosis, participants will be tested conventional method including Xpert TB/RIF assay, and new diagnostic technique using homobifunctionalImidoesters compounds.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are suspected with pulmonary tuberculosis, tuberculosis meningitis, tuberculosis peritonitis, tuberculosis pleurisy

Exclusion Criteria:

* Under 18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of new diagnostic technique | Time Frame: An average of 2 year
  sensitivity and specificity of new test

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, Songpa, South Korea

IPD SHARING:
Plan to Share IPD: No